CLINICAL TRIAL: NCT01359930
Title: Phase 1 Study of Interactions Between Oral Naltrexone and Bupropion and Intravenous Methamphetamine in Methamphetamine Experienced Volunteers
Brief Title: Phase 1 Naltrexone-Bupropion-Methamphetamine Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NaltrexoneBupropion-Ph1A-met
Record Dates: First submitted 2011-05-18; First posted 2011-05-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2013-07

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Naltrexone and Bupropion SR (Active Comparator)
  Interventions: Drug: Naltrexone and Bupropion SR
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — matching placebo
  Arms: Placebo
Drug: Naltrexone and Bupropion SR — 25mg bid/day (NX) 200mg bid/day (BUP)
  Arms: Naltrexone and Bupropion SR

SUMMARY:
The study is to primarily measure safety and interactions between oral doses of Naltrexone/Bupropion and i.v. Methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* Are MA experienced but not dependent, males or females aged 21-to-50 years.
* Reported use of MA during the past six months without experiencing an adverse consequence plus a life time MA or amphetamine use history of at least four occasions of use.
* Have a body mass index (BMI) between 18 and 30.
* Are willing and able to give written consent.
* Are not currently a subject (including still in the follow-up period) of another drug research study.
* Have no medical contraindications determined by the following: an adequate medical history, a physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
* Have a negative drug test for barbiturates, benzodiazepines, opiates, cocaine, amphetamines and ethanol at the time of hospital admission (Day 0).
* Are females who have a negative pregnancy test at hospital admission.
* Are of either non-childbearing (tubal ligation or total hysterectomy) or of childbearing potential using one or more of the following barrier methods of contraception: male or female condoms (with/without spermicide), diaphragm (with spermicide) and/or copper containing intrauterine device (with/without spermicide). No other contraceptives are acceptable.

Exclusion Criteria:

* Please contact site for more information

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular System Effects | daily during the 10 day treatment period
  Heart rate, blood pressure, ECGs,and monitoring adverse events
Number of subjects with adverse events | Day 0 through Day 10

SECONDARY OUTCOMES:
Plasma concentrations obtained at specific timepoints | daily during the 10 day treatment period
  * PK of IV (meth) and its metabolites before and during Naltrexone/BUP exposure
  * PK of bupropion, naltrexone and their metabolites
Assessment of Vital Signs and Clinical Chemistries | Daily during the 10 day treatment period
  Respiration rate and clinical laboratory measures
Cognitive Assessments as reported by the subject | Dailly during the 10 day treatment period
  Subject reported effects measured with VAS, BSCS, and POMS

CONTACTS AND LOCATIONS:
Locations (1):
- Langley Porter Psychiatric Institute, San Francisco, California, United States